CLINICAL TRIAL: NCT02477930
Title: Prospective Registry The Treatment Of Upper And Lower Intestinal Anastomotic Leaks And Perforations
Brief Title: Endosponge Vacuum Therapy (E-VAC) Registry of Intestinal Anastomotic Leaks and Perforations
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 014-263
Record Dates: First submitted 2015-06-19; First posted 2015-06-23 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Intestinal Anastomotic Leak; Intestinal Perforations
MeSH Terms: conditions — Intestinal Perforation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No interventions are done — No intervention is done. This is a registry study.

SUMMARY:
The purpose of this registry is to collect data on the clinical use of endoluminal vacuum (E-Vac) therapy to treat both upper and lower intestinal leaks and perforations.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing E-Vac Therapy
* Age > 17 years

Exclusion Criteria:

* 17 years of age or younger
* Undergone an E-Vac placement > 14 days before consenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's with upper and lower intestinal anastomotic leaks and perforations who are referred for E-Vac therapy or are the primary patients of Dr. Leeds and Dr. Burdick will be invited to participate in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
In-Hospital survival-rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Leeds, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States